CLINICAL TRIAL: NCT06713473
Title: Reducing Self-Dehumanization to Examine the Effects on Oxytocin and Suicide Risk
Brief Title: Reducing Self-Dehumanization to Examine Oxytocin and Suicide Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Thomas Joiner, Robert O. Lawton Distinguished Professor of Psychology, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FP00007283-2
Record Dates: First submitted 2024-11-26; First posted 2024-12-03 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Rehumanization Intervention; Control Intervention
Keywords: self-dehumanization; suicidal ideation; oxytocin
MeSH Terms: conditions — Suicidal Ideation | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehumanized Intervention (Experimental): This self-rehumanization intervention will involve a set of multi-sensory activities (i.e., reading, writing, and speaking) to prompt body and soul awareness, agency, connection, and creativity.
  Interventions: Other: Rehumanized Intervention; Diagnostic Test: Clinical Interview; Other: Self-Report Measures; Other: Blood Draw
- Control Intervention (Active Comparator): Control Intervention about political attitudes
  Interventions: Other: Control Intervention; Diagnostic Test: Clinical Interview; Other: Self-Report Measures; Other: Blood Draw

INTERVENTIONS:
Other: Rehumanized Intervention — Participants will:
  1. be provided with a lay summary of an ostensible research article that used quantitative and qualitative data to capture the experiences of feeling "less than human" and mechanisms for reclaiming human identity. The summary will reveal general themes of humanness based on participant responses including body and soul awareness, agency, connection, and creativity.
  1. write a 30-minute reflective essay on "how did the rehumanization efforts described in the survey make people feel more human?" where they will be encouraged to use examples from their own lives
  2. asked to create videos based on the insights shared in the essays. The researchers will explain, "We would like to record you reading your essay on camera. We believe it would be especially impactful for clinicians developing these interventions to hear directly from someone who has recently navigated similar experiences."
  Arms: Rehumanized Intervention
Other: Control Intervention — Participants will:
  1. be provided with a lay summary of an ostensible research article that used quantitative and qualitative data to capture the experiences of political attitudes and routes to political sophistication. The summary will reveal general themes of political sophistication based on participant responses including gathering information through diverse news outlets, analyzing policy and legislation, and participation in civic engagement
  1. write a 30-minute reflective essay on ""how did the political efforts described in the survey refine political attitudes?" where they will be encouraged to use examples from their own lives
  2. asked to create videos based on the insights shared in the essays. The researchers will explain, "We plan to take excerpts of what you write here and share it with future voters to aid in developing political attitudes."
  Arms: Control Intervention
Diagnostic Test: Clinical Interview — Self-Injurious Thoughts and Behaviors Interview-Short Form (SITBI-SF). Participants will complete an in-person interview featuring 72-items about their history of self-injury and suicidal behaviors. This interview includes 6 yes/no style questions about suicidal thoughts, suicidal plans, suicidal gestures, suicidal attempts, nonsuicidal self-injury thoughts, and nonsuicidal self-injury. Each category that is endorsed, across the lifetime, has follow up questions surrounding times, duration, intensity, severity, type, and if medical attention was sought. This interview has sound psychometric properties.
Other: Self-Report Measures — Depressive Symptom Index - Suicidality Subscale (DSI-SS). Patient Health Questionnaire-8 (PHQ-8). Interpersonal Needs Questionnaire (INQ). Self-Dehumanization Scale (SDS).
Other: Blood Draw — Five milliliters of blood will be drawn before and after study interventions for the quantification of plasma oxytocin concentrations by certified phlebotomists. Samples will be collected into chilled EDTA tubes, inverted ten times to mix with anticoagulants, and centrifuged at 1600g for 15 minutes at 4˚C. Cleared plasma will be aliquoted into cryotubes and stored at -80˚C. Consistent with expert recommendations, oxytocin levels will be obtained from the samples diluted 1:4 (i.e., oxytocin can be discarded through plasma proteins when incorporating an extraction step before conducting the enzyme-linked immunosorbent assay [ELISA]). Second, to buffer against contrasting concerns, an aliquot of each sample will be analyzed for test-retest purposes. Oxytocin concentrations will be measured using a validated commercially available and sensitive ELISA neurophysin kit (Abcam).

SUMMARY:
The goal of this experiment is to further determine if self-dehumanization is a novel risk factor for suicide. This study will reduce self-dehumanization using a novel re-humanization condition and compare this group to a control group to analyze the pathway between higher perceptions of self-dehumanization, suicidal ideation, and changes in oxytocin concentrations.

It is hypothesized that participants randomly assigned to the re-humanized condition will exhibit decreases in suicidal ideation and increases in oxytocin concentrations as compared to the control condition, which will not display significant changes. Further, we will explore if the magnitude of the oxytocin response will partially mediate the change in suicidal ideation.

DETAILED DESCRIPTION:
Purpose: Humans are inherently social beings, and the need for belonging and connection is fundamental. Severe perceptions of social exclusion, non-belonging, and isolation can result in significant psychological harm, including suicide, which claims nearly 50,000 lives annually in the U.S. and affects over 13 million individuals through suicidal ideation (SI). A key predictor of SI, thwarted belongingness, arises from feelings of exclusion and non-belonging, yet more specificity is needed to identify the types of non-belonging that contribute most to suicide risk. Self-dehumanization-a perception of oneself as less than human-emerges as a promising factor in understanding and mitigating SI, with empirical evidence linking it to anxiety, depression, suicidal ideation, and social withdrawal. Preliminary research suggests that self-dehumanization is influenced by neurobiological processes, particularly oxytocin, a hormone critical to social connectedness and self-perception. Low oxytocin levels have been linked to self-dehumanization, reduced social reengagement, and heightened suicide risk, highlighting its potential as a target for intervention. Building on these insights, this study will experimentally induce and reduce self-dehumanization to examine its effects on SI and oxytocin levels. Thus, this study will use a self-dehumanization induction to analyze its impact on SI and oxytocin. Findings will provide a novel framework for integrating psychotherapeutic and neurobiological strategies into suicide prevention efforts.

Research Design/Method: The present study will utilize an experimental design with two groups, an experimental re-humanized group and a comparison control group.

Procedure: All interested participants will be instructed to fill out the screening survey to determine fit. Eligible participants will be invited to complete the study visit in person. Following consent, participants will complete a pre-induction fasted blood draw of 5 milliliters (i.e., approximately a tablespoon of blood). Next, participants will complete the Self-Injurious Thoughts and Behaviors-Short Form interview with the experimenter and a battery of randomized self-report assessments. After completion, eligible participants will then be randomly categorized into the re-humanization intervention or the control intervention. Following this, they will undergo a post-intervention 5 milliliter fasted blood draw. They will then complete a post-induction battery of self-report measures (see Materials). Participants will be queried for any changes in suicide risk and any current suicidal ideation and intent and will receive appropriate interventions (e.g., means safety counseling, safety planning). Upon completion participants will be compensated and provided mental health resources (e.g., the National Suicide Prevention Lifeline). Participants will be contacted one month later to fill out a brief battery of self-report measures. The appointment is expected to take approximately 2 hours to complete.

Data Analyses: All results will be analyzed in R. First, descriptive statistics and zero-order bivariate correlation analyses will be assessed. For this study, repeated measures analysis of covariance (ANCOVAs) will be used to examine group differences (i.e., the active re-humanized condition and control condition) in changes in oxytocin levels, self-dehumanization scores, and suicidal ideation, controlling for social isolation (i.e., thwarted belongingness, a factor of the Interpersonal Needs Questionnaire). Post-hoc pairwise comparisons will be conducted if the omnibus test indicates statistically significant effects. Following this, exploratory analyses will be conducted to assess if oxytocin partially mediates the relationship between self-dehumanization pre-experimental manipulation and suicide risk post-experimental manipulation (controlling for suicide risk at pre-experimental manipulation) through bootstrapped mediation procedures (i.e., 10,000 samples using the mediation and lavaan packages in R).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 40
* Biological females will be screened to ensure that they have a regular menstrual cycle with a length of 26-30 days and will be scheduled according to their cycle (see Research Strategy for details).
* At least a moderate level of self-dehumanization (i.e., a sum score of 12 or greater out of a possible score of 28) and current suicidal ideation

Exclusion Criteria:

* Participation in the Self-Dehumanized Study by this study team
* A phobia of needles (i.e., trypanophobia)
* Any medical conditions precluding them from engaging in a 10-hour fast (consumption of water is allowed and encouraged)
* Life-threatening suicide risk which would result in taking appropriate steps to ensure safety of the individual (e.g., hospitalization) A psychosis-related diagnosis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change in Suicidal Ideation | This measure will be collected at Baseline and after the experiment (approximately 30 minutes later). Then, suicidal ideation will be collected again 1 month later.
  Suicidal Ideation will be measured using the Depressive Symptom Index-Suicidality Subscale (DSI-SS) where the scores range from 0-12 and higher scores indicate higher levels of suicidal ideation. These analyses will control for Baseline suicidal ideation and the thwarted belongingness sub-scale from the Interpersonal Needs Questionnaire where thwarted belongingness scores range from 1-56 and higher scores indicate greater perceptions of thwarted belongingness.
Change in Oxytocin Levels | This measure will be collected at Baseline and after the experiment (approximately 30 minutes later).
  Five milliliters of blood will be drawn before and after study interventions for the quantification of plasma oxytocin concentrations by certified phlebotomists (including the PI, who is already certified and currently collecting samples for a T-32 supported project). Samples will be collected into chilled EDTA tubes, inverted ten times to mix with anticoagulants, and centrifuged at 1600g for 15 minutes at 4˚C. Cleared plasma will be aliquoted into cryotubes and stored at -80˚C. Consistent with expert recommendations, oxytocin levels will be obtained from the samples diluted 1:4 (i.e., oxytocin can be discarded through plasma proteins when incorporating an extraction step before conducting the enzyme-linked immunosorbent assay [ELISA]). Second, to buffer against contrasting concerns, an aliquot of each sample will be analyzed for test-retest purposes. Oxytocin concentrations will be measured using a validated commercially available and sensitive ELISA neurophysin kit (Abcam).

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD de-identified demographic, self-report, and neurobiological (i.e., oxytocin) data may be shared. Data will not be shared if the participant denies to share their data. Data will be accessible by contacting the Central Contact Person of the study: Morgan Robison (mrobison@psy.fsu.edu). If data are uploaded to a public repository, the external link will be made available here.

REFERENCES:
- [Background] Robison M, Jeon ME, Udupa NS, Potter M, Robertson L, Joiner T. The Self-Dehumanization Scale: Three Studies on Its Development and Validation. J Pers Assess. 2025 Jan-Feb;107(1):41-57. doi: 10.1080/00223891.2024.2367543. Epub 2024 Jun 28. PMID 38940620
- [Background] Robison M, Abderhalden FP, Joiner TE. Dehumanization and the Association With Nonsuicidal Self-Injury and Suicidal Ideation in an Incarcerated Population. Crisis. 2024 Jul;45(4):287-293. doi: 10.1027/0227-5910/a000952. Epub 2024 Mar 5. PMID 38441129